CLINICAL TRIAL: NCT04991857
Title: The Effects and Cost-effectiveness of a Technology-based Family-centered Empowerment (T-FAME) Program on Health and Health Service Utilization Outcomes of Post-discharged Patients With Advanced Heart Failure: A Sequential Mixed Method Study
Brief Title: Technology-based Family-centered Empowerment Program for Heart Failure (T-FAME-HF)
Acronym: T-FAME-HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: T-FAME-HF
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Telerehabilitation; Self Care; Empowerment; Disease Management
Keywords: Heart Failure; Telerehabilitation; Self Care; Empowerment; Disease Management
MeSH Terms: conditions — Heart Failure; Empowerment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It is a single-blind study. A research assistant (RA1) will identify eligible patients (participants) by record review, invite their participation and obtain their informed consent. After recruiting the participants, simple randomization will be conducted using a computer-generated sequence by 2-stage block randomization (block size of 8, 10 or 12) in 1:1 allocation ratio for the subjects to receive either the T-FAME-HF or HF education program. Single blinding is maintained by using the another research assistant (RA2), who has no information about group assignment, to collect the post-test self-reported data on outcome variables (i.e. self-care, HRQL and family functioning) via telephone interview.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The technology-based family-centered empowerment program for heart failure (T-FAME-HF) (Experimental): The T-FAME-HF is a 16-week program adopts a hybrid approach to combine nurse-led home visits, an Apps, tele-care and optimized family support to enhance post-discharge disease management, disease monitoring, and patients' access to the nurse, and telephone visits. The Program includes 3 four-week phases, which followed by 2 bi-weekly telephone visits. Each phase is designated with a specified goal of care to guide the disease management activities. Commenced with the home visit by the team nurse for each phase, patients' condition and self-care will be assessed. A goal-setting approach will be used to enhance disease monitoring, symptom recognition and response, and treatment compliance. A mobile apps (T-FAME) will be installed in participants' smart-phone and supports the prescribed actions for goal attainment.
  Interventions: Other: T-FAME-HF
- Control group - HF education program (Active Comparator): For patients assigned to the control arm will receive HF education program, the care dyad will receive a 16-week HF education program that comprises a home visit by another team nurse, five bi-weekly online training on self-care through videos on Whatapps/ WeChat with two subsequent telephone follow-up.
  Interventions: Other: Control group - HF education program

INTERVENTIONS:
Other: T-FAME-HF — 16-week program adopts a hybrid approach to combine nurse-led home visits, an Apps, tele-care and optimized family support to enhance post-discharge disease management, disease monitoring, and patients' access to the nurse, and telephone visits
  Arms: The technology-based family-centered empowerment program for heart failure (T-FAME-HF)
Other: Control group - HF education program — For patients assigned to the control arm will receive HF education program, the care dyad will receive a 16-week HF education program that comprises a home visit by the team nurse, five bi-weekly online training on self-care through videos on Whatapps/ WeChat with two subsequent telephone follow-up.
  Arms: Control group - HF education program

SUMMARY:
Heart failure (HF) is a complex clinical syndrome characterized by inefficient myocardial pumping with signs of pulmonary and systemic congestion. Its progressively deteriorating trajectory punctuated by episodes of acute disease decompensation, not only compromises patients' health-related quality of life (HRQL), but also causes a hospitalization epidemic. Indeed, this clinical cohort is characterized by exceptionally high readmission rate of 25% and 50% within 4 weeks and 6 months, respectively, with ineffective self-care being as the most prominent modifiable risk factor. Effective transitional care is crucial to enhance the patient outcomes and control the economic impact. However, the concerned service in Hong Kong is rather under-developed due to the human resource burden and inadequate integration of the primary and tertiary healthcare systems. In fact, family support is of utmost important to support the HF patients in the post-discharge period. Together with the advance in E-health intervention, this study aims to evaluate the effects and cost-effectiveness of a technology-based family-centered empowerment program (T-FAME) to enhance the self-care and post-discharge outcomes of this clinical cohort.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effects of the technology-based family-centered empowerment program for heart failure (T-FAME-HF) on hospital readmission, mortality, event-free survival, HF-related self-care, family functioning and HRQL among patients admitted with HF. The study targets to recruit 270 participants in local hospitals in total.

The T-FAME-HF is a 16-week program adopts a hybrid approach to combine nurse-led home visits, an Apps, tele-care and optimized family support to enhance the post-discharge disease management, disease monitoring, and patients' access to the nurse, and telephone visits. The Program includes 3 four-week phases (1st - 4th; 5th - 8th; 9th - 12th week), which followed by 2 bi-weekly telephone visits. Each phase is designated with a specified goal of care to guide the disease management activities. Commenced with the home visit by the team nurse for each phase, patients' condition and self-care will be assessed. A goal-setting approach will be used to enhance disease monitoring, symptom recognition and response, and treatment compliance. The T-FAME Apps supports the prescribed actions for goal attainment by facilitating: i) BP and symptom monitoring with provision of corresponding health advice, ii) nurses' disease monitoring, iii) video-based training on knowledge and skills, iv) easy access to nurse through real-time chatroom, and v) weather and air quality alert. A blood pressure monitor device will be provided to support the health monitoring. After the 3rd phase, the nurse will monitor goal-attainment via tele-care.

For patients who assigned into the control group will receive a HF education program, the care dyad will receive a 16-week HF education program that comprises a home visit by another team nurse, five bi-weekly online training on self-care through videos on Whatapps/ WeChat with two subsequent telephone follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients consecutively admitted with a primary diagnosis of HF according to the Framingham criteria will be recruited. Eligible patients will be Chinese over 18 year-old, to be discharged home and living with family, patient/ family are using Smart Phone, and be communicable with the research team.

Exclusion Criteria:

* Those who are awaiting revascularization, cardiac resynchronization or heart transplant, and those with end-stage renal disease relying on hemodialysis rather than HF medications, to regulate fluid volume, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2021-09-19 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Minnesota Living with Heart Failure (MLHF) questionnaire | Baseline
  Measure the disease-specific health-related quality of life (HRQL). There are 21 items and each item is rated from 0 to 5, with higher scores indicating worse outcome.
Minnesota Living with Heart Failure (MLHF) questionnaire | 8th week
  Measure the disease-specific health-related quality of life (HRQL). There are 21 items and each item is rated from 0 to 5, with higher scores indicating worse outcome.
Minnesota Living with Heart Failure (MLHF) questionnaire | 16th week
  Measure the disease-specific health-related quality of life (HRQL). There are 21 items and each item is rated from 0 to 5, with higher scores indicating worse outcome.
Minnesota Living with Heart Failure (MLHF) questionnaire | 24th week
  Measure the disease-specific health-related quality of life (HRQL). There are 21 items and each item is rated from 0 to 5, with higher scores indicating worse outcome.
Minnesota Living with Heart Failure (MLHF) questionnaire | 32th week
  Measure the disease-specific health-related quality of life (HRQL). There are 21 items and each item is rated from 0 to 5, with higher scores indicating worse outcome.

SECONDARY OUTCOMES:
Self-Care Heart Failure Index (SCHFI, v.7.2) | Baseline
  Measure the self-care maintenance, self-care management, and symptom perception of the HF patients. There are 28 questions are rated from 1 to 5, and one question are rated from 0 to 5. The three subscale scores are transformed to 0-100, with higher scores indicating better self-care attributes.
Self-Care Heart Failure Index (SCHFI, v.7.2) | 8th week
  Measure the self-care maintenance, self-care management, and symptom perception of the HF patients. There are 28 questions are rated from 1 to 5, and one question are rated from 0 to 5. The three subscale scores are transformed to 0-100, with higher scores indicating better self-care attributes.
Self-Care Heart Failure Index (SCHFI, v.7.2) | 16th week
  Measure the self-care maintenance, self-care management, and symptom perception of the HF patients. There are 28 questions are rated from 1 to 5, and one question are rated from 0 to 5. The three subscale scores are transformed to 0-100, with higher scores indicating better self-care attributes.
Self-Care Heart Failure Index (SCHFI, v.7.2) | 24th week
  Measure the self-care maintenance, self-care management, and symptom perception of the HF patients. There are 28 questions are rated from 1 to 5, and one question are rated from 0 to 5. The three subscale scores are transformed to 0-100, with higher scores indicating better self-care attributes.
Self-Care Heart Failure Index (SCHFI, v.7.2) | 32th week
  Measure the self-care maintenance, self-care management, and symptom perception of the HF patients. There are 28 questions are rated from 1 to 5, and one question are rated from 0 to 5. The three subscale scores are transformed to 0-100, with higher scores indicating better self-care attributes.
Self-Care Self-Efficacy Scale (SCSE) | Baseline
  Evaluate the confidence level of patients with chronic disease on their self-care self-efficacy. There are 10 items and each item is rated from 1 (not confident) to 5 (extremely confident), with higher scores indicating better self-care attributes.
Self-Care Self-Efficacy Scale (SCSE) | 8th week
  Evaluate the confidence level of patients with chronic disease on their self-care self-efficacy. There are 10 items and each item is rated from 1 (not confident) to 5 (extremely confident), with higher scores indicating better self-care attributes.
Self-Care Self-Efficacy Scale (SCSE) | 16th week
  Evaluate the confidence level of patients with chronic disease on their self-care self-efficacy. There are 10 items and each item is rated from 1 (not confident) to 5 (extremely confident), with higher scores indicating better self-care attributes.
Self-Care Self-Efficacy Scale (SCSE) | 24th week
  Evaluate the confidence level of patients with chronic disease on their self-care self-efficacy. There are 10 items and each item is rated from 1 (not confident) to 5 (extremely confident), with higher scores indicating better self-care attributes.
Self-Care Self-Efficacy Scale (SCSE) | 32th week
  Evaluate the confidence level of patients with chronic disease on their self-care self-efficacy. There are 10 items and each item is rated from 1 (not confident) to 5 (extremely confident), with higher scores indicating better self-care attributes.
The EuroQoL-5-D instruments | Baseline
  Assess the health-related quality of life of the care dyads and to generate the utility score for cost-effective analysis. It consists of two parts, with the first part to assess the health status on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a 5-level (no problems, slight problems , moderate problems, severe problems and unable to) response set, with "unable to" levels mean a worse situation. The second part as a 0-100 scores VAS to measure perceived health, higher scores mean a better outcome.
The EuroQoL-5-D instruments | 8th week
  Assess the health-related quality of life of the care dyads and to generate the utility score for cost-effective analysis. It consists of two parts, with the first part to assess the health status on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a 5-level (1 to 5) response set, with higher levels mean a worse situation. The second part as a 0-100 scores VAS to measure perceived health, higher scores mean a better outcome.
The EuroQoL-5-D instruments | 16th week
  Assess the health-related quality of life of the care dyads and to generate the utility score for cost-effective analysis. It consists of two parts, with the first part to assess the health status on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a 5-level (no problems, slight problems , moderate problems, severe problems and unable to) response set, with "unable to" levels mean a worse situation. The second part as a 0-100 scores VAS to measure perceived health, higher scores mean a better outcome.
The EuroQoL-5-D instruments | 24th week
  Assess the health-related quality of life of the care dyads and to generate the utility score for cost-effective analysis. It consists of two parts, with the first part to assess the health status on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a 5-level (no problems, slight problems , moderate problems, severe problems and unable to) response set, with "unable to" levels mean a worse situation. The second part as a 0-100 scores VAS to measure perceived health, higher scores mean a better outcome.
The EuroQoL-5-D instruments | 32th week
  Assess the health-related quality of life of the care dyads and to generate the utility score for cost-effective analysis. It consists of two parts, with the first part to assess the health status on mobility, self-care, usual activities, pain/discomfort, and anxiety/depression using a 5-level (no problems, slight problems , moderate problems, severe problems and unable to) response set, with "unable to" levels mean a worse situation. The second part as a 0-100 scores VAS to measure perceived health, higher scores mean a better outcome.
Family Assessment Device Questionnaire - Global Family Function Subscale | Baseline
  Measure the patients' perception of the overall function of the family in supporting the disease management. Each item is rated from one to four (strongly agree, agree, disagree and strongly disagree), higher scores mean a worse outcome.
Family Assessment Device Questionnaire - Global Family Function Subscale | 8th week
  Measure the patients' perception of the overall function of the family in supporting the disease management. Each item is rated from one to four (strongly agree, agree, disagree and strongly disagree), higher scores mean a worse outcome.
Family Assessment Device Questionnaire - Global Family Function Subscale | 16th week
  Measure the patients' perception of the overall function of the family in supporting the disease management. Each item is rated from one to four (strongly agree, agree, disagree and strongly disagree), higher scores mean a worse outcome.
Family Assessment Device Questionnaire - Global Family Function Subscale | 24th week
  Measure the patients' perception of the overall function of the family in supporting the disease management. Each item is rated from one to four (strongly agree, agree, disagree and strongly disagree), higher scores mean a worse outcome.
Family Assessment Device Questionnaire - Global Family Function Subscale | 32th week
  Measure the patients' perception of the overall function of the family in supporting the disease management. Each item is rated from one to four (strongly agree, agree, disagree and strongly disagree), higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Sau Fung YU, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Medicine, PoK Oi Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Only study investigators and research assistants involved in the study will have access to the data.

REFERENCES:
- [Result] Murray SA, Kendall M, Boyd K, Sheikh A. Illness trajectories and palliative care. BMJ. 2005 Apr 30;330(7498):1007-11. doi: 10.1136/bmj.330.7498.1007. No abstract available. PMID 15860828
- [Result] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Result] Coleman EA, Boult C; American Geriatrics Society Health Care Systems Committee. Improving the quality of transitional care for persons with complex care needs. J Am Geriatr Soc. 2003 Apr;51(4):556-7. doi: 10.1046/j.1532-5415.2003.51186.x. No abstract available. PMID 12657079
- [Result] Vedel I, Khanassov V. Transitional Care for Patients With Congestive Heart Failure: A Systematic Review and Meta-Analysis. Ann Fam Med. 2015 Nov;13(6):562-71. doi: 10.1370/afm.1844. PMID 26553896
- [Result] Stamp KD, Prasun M, Lee CS, Jaarsma T, Piano MR, Albert NM. Nursing research in heart failure care: a position statement of the american association of heart failure nurses (AAHFN). Heart Lung. 2018 Mar-Apr;47(2):169-175. doi: 10.1016/j.hrtlng.2018.01.003. Epub 2018 Feb 15. PMID 29397988
- [Result] Griffiths SM, Lee JP. Developing primary care in Hong Kong: evidence into practice and the development of reference frameworks. Hong Kong Med J. 2012 Oct;18(5):429-34. PMID 23018072
- [Result] Smith J, Ali P, Birks Y, Curtis P, Fairbrother H, Kirk S, Saltiel D, Thompson J, Swallow V. Umbrella review of family-focused care interventions supporting families where a family member has a long-term condition. J Adv Nurs. 2020 Aug;76(8):1911-1923. doi: 10.1111/jan.14367. Epub 2020 Apr 15. PMID 32215957
- [Result] Deek H, Hamilton S, Brown N, Inglis SC, Digiacomo M, Newton PJ, Noureddine S, MacDonald PS, Davidson PM; FAMILY Project Investigators. Family-centred approaches to healthcare interventions in chronic diseases in adults: a quantitative systematic review. J Adv Nurs. 2016 May;72(5):968-79. doi: 10.1111/jan.12885. Epub 2016 Jan 10. PMID 26751971
- [Result] Ostergaard B, Mahrer-Imhof R, Wagner L, Barington T, Videbaek L, Lauridsen J. Effect of family nursing therapeutic conversations on health-related quality of life, self-care and depression among outpatients with heart failure: A randomized multi-centre trial. Patient Educ Couns. 2018 Aug;101(8):1385-1393. doi: 10.1016/j.pec.2018.03.006. Epub 2018 Mar 7. PMID 29567335
- [Result] Ho KK, Anderson KM, Kannel WB, Grossman W, Levy D. Survival after the onset of congestive heart failure in Framingham Heart Study subjects. Circulation. 1993 Jul;88(1):107-15. doi: 10.1161/01.cir.88.1.107. PMID 8319323
- [Result] Yu DS, Lee DT, Stewart S, Thompson DR, Choi KC, Yu CM. Effect of Nurse-Implemented Transitional Care for Chinese Individuals with Chronic Heart Failure in Hong Kong: A Randomized Controlled Trial. J Am Geriatr Soc. 2015 Aug;63(8):1583-93. doi: 10.1111/jgs.13533. PMID 26289684
- [Result] Riegel B, Barbaranelli C, Carlson B, Sethares KA, Daus M, Moser DK, Miller J, Osokpo OH, Lee S, Brown S, Vellone E. Psychometric Testing of the Revised Self-Care of Heart Failure Index. J Cardiovasc Nurs. 2019 Mar/Apr;34(2):183-192. doi: 10.1097/JCN.0000000000000543. PMID 30303894
- [Result] Yu DS, De Maria M, Barbaranelli C, Vellone E, Matarese M, Ausili D, Rejane RE, Osokpo OH, Riegel B. Cross-cultural applicability of the Self-Care Self-Efficacy Scale in a multi-national study. J Adv Nurs. 2021 Feb;77(2):681-692. doi: 10.1111/jan.14617. Epub 2020 Dec 9. PMID 33295675
- [Result] Riegel B, Lee CS, Dickson VV, Carlson B. An update on the self-care of heart failure index. J Cardiovasc Nurs. 2009 Nov-Dec;24(6):485-97. doi: 10.1097/JCN.0b013e3181b4baa0. PMID 19786884
- [Result] Yu DSF, Li PWC, Yue SCS, Wong J, Yan B, Tsang KK, Choi KC. The effects and cost-effectiveness of an empowerment-based self-care programme in patients with chronic heart failure: A study protocol. J Adv Nurs. 2019 Dec;75(12):3740-3748. doi: 10.1111/jan.14162. Epub 2019 Aug 27. PMID 31350765
- [Result] Ho CC, Clochesy JM, Madigan E, Liu CC. Psychometric evaluation of the Chinese version of the Minnesota Living with Heart Failure Questionnaire. Nurs Res. 2007 Nov-Dec;56(6):441-8. doi: 10.1097/01.NNR.0000299849.21935.c4. PMID 18004191
- [Result] Buchholz I, Janssen MF, Kohlmann T, Feng YS. A Systematic Review of Studies Comparing the Measurement Properties of the Three-Level and Five-Level Versions of the EQ-5D. Pharmacoeconomics. 2018 Jun;36(6):645-661. doi: 10.1007/s40273-018-0642-5. PMID 29572719
- [Result] Cheung PWH, Wong CKH, Samartzis D, Luk KDK, Lam CLK, Cheung KMC, Cheung JPY. Psychometric validation of the EuroQoL 5-Dimension 5-Level (EQ-5D-5L) in Chinese patients with adolescent idiopathic scoliosis. Scoliosis Spinal Disord. 2016 Aug 4;11:19. doi: 10.1186/s13013-016-0083-x. eCollection 2016. PMID 27525314
- [Result] Stamp KD, Dunbar SB, Clark PC, Reilly CM, Gary RA, Higgins M, Ryan RM. Family partner intervention influences self-care confidence and treatment self-regulation in patients with heart failure. Eur J Cardiovasc Nurs. 2016 Aug;15(5):317-27. doi: 10.1177/1474515115572047. Epub 2015 Feb 11. PMID 25673525
- [Result] Chen S, Zheng S, Wang X, Zhang X, Fa T, Fu L, Zang X, Zhao Y. Linguistic and Psychometric Validation of the Chinese Version of the Control Attitudes Scale-Revised in Patients With Chronic Heart Failure. J Cardiovasc Nurs. 2021 Jul-Aug 01;36(4):349-356. doi: 10.1097/JCN.0000000000000705. PMID 32472800
- [Result] Zou G. A modified poisson regression approach to prospective studies with binary data. Am J Epidemiol. 2004 Apr 1;159(7):702-6. doi: 10.1093/aje/kwh090. PMID 15033648
- [Result] Liu GG, Wu H, Li M, Gao C, Luo N. Chinese time trade-off values for EQ-5D health states. Value Health. 2014 Jul;17(5):597-604. doi: 10.1016/j.jval.2014.05.007. Epub 2014 Jul 23. PMID 25128053
- [Result] Thompson SG, Barber JA. How should cost data in pragmatic randomised trials be analysed? BMJ. 2000 Apr 29;320(7243):1197-200. doi: 10.1136/bmj.320.7243.1197. No abstract available. PMID 10784550
- [Result] Fenwick E, O'Brien BJ, Briggs A. Cost-effectiveness acceptability curves--facts, fallacies and frequently asked questions. Health Econ. 2004 May;13(5):405-15. doi: 10.1002/hec.903. PMID 15127421
- See also: Hospital Authority. Hospital Authority Statistical Report 2011/ 2012. Hong Kong: Hong Kong Hospital Authority; 2013. — https://www3.ha.org.hk/data/HAStatistics/DownloadReport/6?isPreview=False

DOCUMENTS (1):
  • Informed Consent Form (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04991857/ICF_000.pdf